CLINICAL TRIAL: NCT05430295
Title: Distance And Intermediate Visual Acuity After Phacoemulsification Using A New Generation Monofocal Intraocular Lens Compared To Standard Monofocal Intraocular Lens
Brief Title: Visual Acuity After Using A New Monofocal Intraocular Lens Compared To Standard Monofocal Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rokaya Emad Radwan, ophthalmology resident, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MS-239-2021
Record Dates: First submitted 2022-04-13; First posted 2022-06-24 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Lenses, Intraocular
Keywords: intraocular lens; intermediate vision; contrast sensitivity; monofocal
MeSH Terms: interventions — Phacoemulsification; Cataract Extraction

STUDY DESIGN:
Intervention Model Description: This is a prospective comparative interventional clinical study,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Eyhance intraocular lens (Active Comparator): 10 patients bilaterally implanted with Eyhance intraocular lens
  Interventions: Procedure: phacoemulsification; Procedure: monofocal intraocular lens implantation
- Tecnis 1 piece intraocular lens (Active Comparator): 10 patients bilaterally implanted with Tecnis 1 piece intraocular lens
  Interventions: Procedure: phacoemulsification; Procedure: monofocal intraocular lens implantation

INTERVENTIONS:
Procedure: phacoemulsification — cataract extraction followed by bilateral implantation of Eyhance intraocular lens in 10 patients and bilateral implantation of Tecnis 1 piece IOL in 10 patients
  Other Names: cataract extraction
Procedure: monofocal intraocular lens implantation — implantation of monofocal intraocular lens in the capsular bag at the end of phacoemulsification surgery

SUMMARY:
This is a prospective comparative interventional clinical study, that took place from January 2021 to November 2021. Twenty patients (20) were enrolled in this study 10 patients in each group. It was designed for comparison of uncorrected and best corrected distance and intermediate vision in patients whom implanted with monofocal Tecnis Eyhance or Tecnis 1-piece IOLs.

DETAILED DESCRIPTION:
Purpose To determine the Uncorrected and best-corrected distance, and intermediate visual acuity in a new innovative monofocal intraocular lens compared with standard monofocal lens.

Methods This is a prospective comparative interventional clinical study, that took place from January 2021 to November 2021. 40 eyes of Twenty patients (20) were enrolled in this study, patients who are candidates for cataract extraction by phacoemulsification were included in this study and underwent thorough preoperative examination and post-operative evaluation at 3 months after the 2nd eye operation, of distance, intermediate, near add, contrast sensitivity and incidence of photic phenomena using a printed questionnaire for evaluating this incidence and binocular defocus curves were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-75 years old undergoing cataract surgery.
* Preoperative corneal astigmatism equal to or less than - 1.00 D.
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures

Exclusion Criteria:

* Visual potential of less than 0.63 due to ocular pathologies.
* Corneal astigmatism over -1.00 D cylinder.
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils, or pupils that do not dilate at least 3.5 mm under mesopic/scotopic conditions).
* Capsule or zonular abnormalities that would affect postoperative centration or tilt of the lens and pseudoexfoliation syndrome.
* Macular degeneration, cystoid macular edema,Diabetic retinopathy, history of uveitis, optic nerve diseases, glaucoma and amblyopia.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Uncorrected and best-corrected distance, and intermediate visual acuity. | 3 months post operative
  Distance visual acuities were examined by ETDRS chart and intermediate and near visual acuity by Jaeger chart at 66 cm and 33 cm respectively.Measured values of the visual acuity were expressed in decimal values and converted to logMAR values.

SECONDARY OUTCOMES:
Contrast sensitivity | 3 months post operative
  Contrast sensitivity was measured using Pelli Robson illuminated chart at 1m

CONTACTS AND LOCATIONS:
Overall Officials: yehia Salaheldin, PhD, Study Director — Cairo University
Locations (1):
- Kasraliany Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
the data of the patients are kept in files with the principal investigator

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/95/NCT05430295/Prot_SAP_001.pdf